CLINICAL TRIAL: NCT06947785
Title: Effectiveness of Combined Neural Mobilization With Manual Myofascial Release for Sciatic Pain Relief
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01004 Anwar Ullah
Record Dates: First submitted 2025-04-07; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Sciatica
Keywords: Neural Mobilization; Myofascial Release; Sciatic Pain
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Neural Mobilization with Manual myofascial Release (Experimental): Combined neural mobilization of Sciatic nerve and manual myofascial release of piriformis and back muscles will be given to this group.
  Interventions: Other: Combined Neural Mobilization with Manual myofascial Release
- Neural Mobilization (Active Comparator): Only neural mobilization of Sciatic nerve will be given to this group.
  Interventions: Other: Neural Mobilization
- Manual Myofascial Release (Active Comparator): Only manual myofascial release of piriformis and back muscles will be given to this group.
  Interventions: Other: Manual Myofascial Release

INTERVENTIONS:
Other: Combined Neural Mobilization with Manual myofascial Release — Combined neural mobilization with manual myofascial release will be provided to each subject.
  Other Names: Neural Mobilization; Manual Myofascial Release
  Arms: Combined Neural Mobilization with Manual myofascial Release
Other: Neural Mobilization — neural mobilization will be provided to each subject.
  Other Names: Combined Neural Mobilization with Manual myofascial Release; Manual Myofascial Release
  Arms: Neural Mobilization
Other: Manual Myofascial Release — Manual myofascial release will be provided to each subject.
  Other Names: Combined Neural Mobilization with Manual myofascial Release; Neural Mobilization
  Arms: Manual Myofascial Release

SUMMARY:
This study will address to evaluate and compare both Neural mobilization and Manual Myofascial Release of piriformis and Lumbar muscles in sciatic pain with the aim of evaluating and identifying the most effective intervention for managing this specific condition, and provide valuable insights into the effectiveness, mechanisms, and practical considerations associated with these interventions, ultimately contributing to evidence based and patient centered care.

DETAILED DESCRIPTION:
MFR is a hands-on technique targeting fascial restrictions that may contribute to pain and reduced mobility. Barnes proposed that releasing fascial adhesions can improve circulation, reduce nerve compression, and enhance tissue flexibility. In a study by Ajimsha et al. , MFR was found to significantly reduce pain and improve physical function in patients with nonspecific low back pain. There is a lack of comparative research assessing the relative efficacy of neural mobilization andMFR in sciatic pain management. While both techniques are rooted in distinct mechanisms neural desensitization versus fascial release they may have overlapping benefits in improving mobility and reducing pain. This study addresses this research gap by directly comparing the two approaches in individuals with sciatic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed unilateral sciatic pain for >3 months.
2. Positive Straight Leg Raise (SLR).

Exclusion Criteria:

- Participants fall in this category would be excluded of the study.

1. Recent spinal surgery or trauma.
2. Neurological deficits or systemic conditions affecting the nervous system.
3. Any other red flags

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | Four Weeks
  A subjective pain assessment tool where patients rate their pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain).
Universal Goniometer | Four Weeks
  Joint range of motion will be measured using a Universal Goniometer in degrees (°). Each joint movement will be assessed individually. The goniometer will be used following standardized procedures as per the American Academy of Orthopaedic Surgeons (AAOS) guidelines. Unit of Measure is degrees.
Patient-Specific Functional Scale | Four Weeks
  The Patient-Specific Functional Scale is a validated patient-reported outcome measure used to assess functional limitations based on activities identified by the patient. Participants will rate their ability to perform 3-5 self-selected activities that are important to them, using an 11-point scale ranging from 0 to 10.
  Minimum score: 0 (indicating the patient is unable to perform the activity)
  Maximum score: 10 (indicating the patient can perform the activity at their prior level with no difficulty)
  Interpretation: Higher scores indicate better functional status.
  The average score across all selected activities will be used for analysis.
SLR (Straight Leg Raise) | Four Weeks
  A clinical test used to assess sciatic nerve irritation or lumbar radiculopathy by raising the extended leg while the patient lies supine.

CONTACTS AND LOCATIONS:
Overall Officials: Amnah Anum, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Malakand, Chakdara, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No